CLINICAL TRIAL: NCT06730750
Title: A Phase 1/2a, Multicenter, Open-label, First in Human Study of BMS-986490 With or Without Bevacizumab in Advanced Solid Tumors
Brief Title: A Study of BMS-986490 With or Without Bevacizumab in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA238-0001; 2024-518421-14 (Other: EU CTR); U1111-1313-7004 (Other: WHO)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Colorectal Cancer (CRC); Non-small Cell Lung cancer (NSCLC); Gastric Cancer (GC)
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A (Experimental)
  Interventions: Drug: BMS-986490
- Part 2A - Colorectal Cancer (CRC) (Experimental)
  Interventions: Drug: BMS-986490
- Part 2A - Non-Small Cell Lung Cancer/Gastric Cancer (NSCLC/GC) (Experimental)
  Interventions: Drug: BMS-986490
- Part 1B (Experimental)
  Interventions: Drug: BMS-986490; Drug: Bevacizumab
- Part 2B (Experimental)
  Interventions: Drug: BMS-986490; Drug: Bevacizumab

INTERVENTIONS:
Drug: BMS-986490 — Specified dose on specified days.
Drug: Bevacizumab — Specified dose on specified days.
  Arms: Part 1B; Part 2B

SUMMARY:
This is a study of BMS-986490 as a monotherapy and in combination with bevacizumab in participants with select advanced solid tumors known to express CEACAM5.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically or cytologically confirmed, advanced, unresectable/metastatic solid tumor measurable by RECIST v1.1.
* CRC: Part 1A, Part 2A-CRC, Part 1B, and Part 2B:

  i) Locally advanced/metastatic, recurrent, or unresectable CRC with adenocarcinoma histology and whose disease has progressed after systemic cancer therapy in the metastatic or adjuvant setting including 5-FU, irinotecan, and/or oxaliplatin (if available and not contraindicated).
* NSCLC: Part 2A-NSCLC/GC, 2L+ NSCLC:

  i) Histologically confirmed NSCLC meeting stage criteria for Stage IIIB, Stage IV, or recurrent disease.

ii) Participants must have received and progressed on or after anti-PD-(L)1 therapy, if available.

- GC: Part 2A-NSCLC/GC, 2L+ GC: i) Participants must have received and then progressed or been intolerant to at least 1 standard treatment regimen in the advanced or metastatic setting (or have progressed within 6 months of adjuvant therapy).

ii) ECOG performance status of 0 or 1.

Exclusion Criteria:

* History of anaphylactic reactions to irinotecan and/or bevacizumab.
* Previously received therapy targeting CEACAM5.
* Grade ≥3 ILD/pneumonitis.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2029-12-09 (Estimated)

PRIMARY OUTCOMES:
Number of participnats with Adverse Events (AEs) | Up to 100 days following discontinuation of dosing
Number of participants with Serious AEs (SAEs) | Up to 100 days following discontinuation of dosing
Number of participants with AEs meeting protocol-defined dose limiting toxicity (DLT) criteria | Up to 28 days after the first treatment of study intervention
Number of participants with AEs leading to discontinuation | Up to 100 days following discontinuation of dosing
Number of deaths | Up to 100 days following discontinuation of dosing

SECONDARY OUTCOMES:
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Approximately 30 Days after Cycle 30, Day 1 (1 Cycle = 21 Days)
Trough observed concentration (Ctrough) | Approximately 30 Days after Cycle 30, Day 1 (1 Cycle = 21 Days)
Maximum observed concentration (Cmax) | Approximately 30 Days after Cycle 30, Day 1 (1 Cycle = 21 Days)
Time of maximum observed concentration (Tmax) | Approximately 30 Days after Cycle 30, Day 1 (1 Cycle = 21 Days)
Total anti-drug antibodies (ADAs) | Approximately 30 Days after Cycle 30, Day 1 (1 Cycle = 21 Days)
Objective Response Rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 assessed by Investigator | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (4):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - START Midwest, Grand Rapids, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
- Tasman Oncology Research, Southport, Queensland, Australia
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06730750.html